CLINICAL TRIAL: NCT07077447
Title: DaBlaCa 23 - The European Collaborative Study on Upper Urinary Tract Urothelial Carcinoma
Brief Title: The Danish Bladder Cancer Group 23 Study - A European Study on Cancer in the Upper Urinary Tract
Acronym: EuroCUT
Status: Recruiting | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Aarhus University Hospital Skejby (Other); Rigshospitalet, Denmark (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: SJ-1085; p-2024-17586 (Other: Region Zealand Research Directory)
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-06

CONDITIONS: Upper Urinary Tract Urothelial Carcinoma
Keywords: UTUC; Upper Urinary Tract Urothelial Carcinoma; Kidney Sparing Surgery; Prospective cohort study; Ureteroscopy; Radical nephroureterectomy; Lynch Syndrome; Endoscopic management of UTUC
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patientens diagnosed with upper urinary tract urothelial carcinoma (UTUC): The study includes all patients diagnosed with upper tract urothelial carcinoma (UTUC) confirmed by histopathology. As a cohort study, it involves no interventions.
  Interventions: Procedure: Kidney sparing surgery for high-risk upper urinary tract urothelial carcinoma

INTERVENTIONS:
Procedure: Kidney sparing surgery for high-risk upper urinary tract urothelial carcinoma — This is an observational cohort study with no direct intervention assigned by the investigators. The study compares two groups of patients in our cohort diagnosed with high-risk pTa upper tract urothelial carcinoma (UTUC), as defined by the European Association of Urology (EAU) guidelines. The "experimental" group includes patients who, due to imperative indications (e.g., solitary kidney, impaired renal function, or comorbidities), undergo kidney-sparing surgery. These patients are compared to a reference group treated with radical nephroureterectomy, which is considered "standard of care".

SUMMARY:
This is a study looking at how patients with a rare type of cancer in the pelvis and ureter of the kidney - called upper urinary tract urothelial carcinoma (UTUC) - is currently treated. The gold standard treatment of UTUC is the complete removal of the kidney, renal pelvis and ureter. The use of kidney-sparing surgery, which preserves the kidney while treating the cancer, was only considered for patients who were too frail to undergo kidney removal, had a solitary functioning kidney, or suffered from severe chronic kidney disease. Since 2018 international guidelines have incorporated kidney sparing surgery for all patients but only offered to patients that have been diagnosed with very low risk tumors to ensure the safety of the patients. The latest update of the UTUC Guidelines from the European Association of Urology has revised the criteria, so that certain features previously classified as high-risk are no longer considered high-risk on their own, provided the tumor otherwise appears benign. Nonetheless, ongoing research is essential to support this evolving approach and to further enhance the guidelines.

Kidney sparing surgery comprise of a strict follow up schedule that often demands supplemental surgeries under general anesthesia, which can cause strain on patients.

Preservation of the kidney is important since a decrease in kidney function can result in increased risk of cardiovascular disease and death.

The main question we want to answer is:

Can more patients with superficial non-invasive UTUC safely be treated with kidney-sparing surgery instead of the more aggressive surgery that removes the entire kidney and ureter without increasing the risk of the cancer coming back and while maintaining quality of life? Furthermore, we are interested in learning more about patients who later develop bladder cancer after treatment of UTUC (intravesical recurrences), the affection of kidney function over time and a subgroup of UTUC patients that are diagnosed with Lynch syndrome (a genetic condition that increases cancer risk and development of UTUC is the third most common cancer) where UTUC presents differently than other patients.

Participants Anyone diagnosed with UTUC can take part in the study. We will collect information from their medical records when they join and again after one, three, five, and ten years. Participants will also be asked to fill out quality-of-life questionnaires at the beginning of entering the study and at one, three and five years.

DETAILED DESCRIPTION:
Detailed description Study Overview and Scientific Rationale Upper urinary tract urothelial carcinoma (UTUC) accounts of 5-10 % of urothelial carcinomas, with an incidence of nearly two cases per 100.000 inhabitants in the western countries. It is estimated that 5-7 % of UTUC are disseminated at time of diagnosis and 60 % are invasive, with a subsequent 5 year overall survival of merely 57% for all UTUC. Age at diagnosis has been increasing over the years, a likely consequence of longer lifespan and better diagnostics, and the mean age at diagnosis is now 70-73 years. Common risk factors are male gender (2:1 ratio to female), smoking and aromatic amines.

Treatments Radical nephroureterectomy (RNU) is considered the gold standard treatment of UTUC, but kidney sparing surgery (KSS) as a treatment option has gained more ground over the years as technology and knowledge about UTUC have improved. Risk stratifications before treatment decisions comprise of imaging of the urinary tract, predominantly CT urography, selective urine cytology and flexible ureteroscopy (fURS). Histopathology assessment of a fURS biopsy can determine the grade of the tumor in more than 90% of cases. However, fURS biopsies are not without limitations, with risk of under staging especially high-grade tumors, and inconclusive biopsies due to small specimen material, since the biopsy forceps usually are 3-4 french in size.

In 2018 the European Association of Urology (EAU) changed its guidelines for low-risk UTUC and now recommend a KSS approach in all patients with low-risk UTUC independent of pre-operative renal function. Low-risk UTUC is defined as: unifocal disease, tumor size < 2 cm, negative for high-grade selected site urine cytology, low-grade fURS biopsy and no invasive aspect on CT.

KSS comprises of three distinct surgical techniques: laser treatment, percutaneous resection, segmental ureter resection (SU) with either end-to-end ureter anastomosis or neoimplantation of the ureter into the bladder. In selected cases patients with high-risk UTUC may also be treated with a KSS approach - ex. in patients with a single kidney, bilateral disease, significant comorbidity or impaired renal function. Some studies indicate that selected high-risk cases diagnosed with low-grade tumors benefit from KSS instead of RNU, regardless of imperative causes. More recently, multifocal low-grade UTUC has been proposed as an intermediate-risk category, rather than being automatically classified as high-risk. This development is reflected in the 2024 EAU UTUC guidelines, which now identify hydroureteronephrosis, multifocality, and tumor size as weak high-risk criteria. Consequently, the presence of one of these features does not automatically preclude KSS if the remaining low-risk criteria are met. It is important to note, that the current evidence base for KSS in UTUC remains limited. The available literature is still developing and largely consists of smaller, retrospective cohort studies.

KSS demands close follow up, as there is a high risk of local recurrence. One study found, that patients treated with RNU had a total of 3.18 procedures performed after a mean follow up of 37.29 months, compared to 8.76 procedures following KSS (follow up 47.81 months), which might impact on the quality of life (QoL). On the other hand, there is evidence that radical nephroureterectomy increases long-term mortality which may be a reflection of the decrease in renal function after RNU. Identification of predictors leading to a postoperative decline in renal function after RNU are mostly retrospective, but the overall consensus suggests that the largest decline is seen in patients with low preoperative eGFR, higher age, postoperative AKI and the absence of hydronephrosis. End-stage CKD can lead to hemodialysis which significantly impairs QoL, and increases morbidity and mortality. The 5-year risk of progression from CKD stage 3 to end-stage kidney disease with the need of dialysis or renal transplant is merely 1.3%. Notably patients with a eGFR of 40 ml/min/1.73m2 have a short life expectancy with a 5-year overall mortality of 25%.

Lynch syndrome Lynch syndrome, also known as hereditary non polyposis colorectal cancer, is caused by the germline mutation of one of four mismatch repair genes (MLH1, MSH2, MSH6 and PMS2) or the EPCAM gene, which can cause inactivation of the MSH2 tumor suppressor gene. These genetic altercations lead to a spectrum of cancers in which UTUC is the third most frequent cancer. Patients with Lynch syndrome have a 14-22 times higher risk of developing UTUC and are diagnosed 10-15 years earlier than the background population. Additionally, UTUC in Lynch patients are more likely to occur in the ureter than in the renal pelvis. In contrast to the general population where men are twice as likely to be diagnosed with UTUC, the gender ratio is 1:1 and there is an increased risk of developing bilateral UTUC. The percentage of patients with UTUC related to Lynch syndrome differs in the literature with rates between 1-20% of Lynch Syndrome related UTUC.

As formerly stated, UTUC is a rare disease and patients with UTUC and Lynch syndrome are even more of a rarity, thus the literature of this corner of UTUC is very scarce. When treating these patients the risk of subsequent contralateral disease must be taken into consideration, thus favoring KSS, but without comprising the oncological outcome for this patient group.

It is recommended that all primary UTUC pathology specimens are screened for the expression of the mismatch repair genes MLH1, MSH2, MSH6 and PMS2 and patients diagnosed with Lynch syndrome follow yearly screenings with an ultrasound, urinary dipstick and cytology.

Intravesical recurrence The risk of intravesical recurrence (IVR) after surgical treatment for UTUC, primarily after RNU, is between 21-50 %, with 82% occurring within the first two years after diagnosis.

IVR is primarily treated with transurethral resection of bladder tumor (TURBT). The follow-up is according to bladder cancer guidelines which are adjusted according to the stage and grade of the tumor. One study presented a mean of 2.3 recurrences/patient. Therefore, follow-up extends for an extra five years beyond the initial diagnosis of IVR. Although studies on treatment for non-muscle invasive bladder cancer may not apply to treatment for IVR after KSS for UTUC, it has been shown that the risk of overall death is 14% higher is patients who have undergone 2-4 TURBTs compared to patients who have only undergone 1.

The role of Mitomycin C (MMC) in preventing IVR is to eradicate any residing tumor cells from the bladder by damaging the DNA of the tumor cells. The ODMID-C trial, a prospective randomized study concluded that a single instillation of MMC after RNU reduces the risk of IVR with absolute risk reduction of 11% and relative risk reduction of 40%.

Rationale and objectives To our knowledge only one multinational prospective UTUC database-study exists, The CROES-UTUC registry, which terminated inclusion in 2019.

The development of treatment options for UTUC has improved over the years. Thus, there is need for further knowledge within the treatment field of UTUC to provide true personalized treatments options to our patients.

EuroCUT is a prospective, multicenter study established to meet the need for feasible, high-volume research capable of generating robust, clinically meaningful data. Originally initiated by Danish Bladder Cancer Group and the Nordic Association of Urology Urothealial Group, the study has now expanded into a broader European collaboration to ensure rapid and achievable patient inclusion.

The collected data will be used to validate the current prediction tools and explore novel tools within the following areas:

1. Prediction on oncological outcomes after RNU or KSS.
2. Prediction of the long-term preservation of renal function after KSS compared to RNU
3. Prediction of IVR after bladder instillation with chemotherapy
4. Prediction of the oncological outcomes for UTUC patients diagnosed with Lynch Syndrome
5. Prediction of patient related outcome measures of patients treated with RNU or KSS.

We hypothesize that we can accommodate these aims and provide further development of the current prediction tools to provide personalized well documented treatment options to our patients.

Study design summary EuroCUT is a prospective, multicenter observational cohort study. No randomization or experimental intervention is applied; clinical management follows routine practice and is determined by the treating physician. Patients are invited to participate in the study at the time of a confirmed histopathology of UTUC.

The study started inclusion in Denmark by November 2025 and expand throughout the European countries by 2026. The study is expected to terminate inclusion by December 2030 and follow up in 2040.

Data are collected at baseline and during follow-up at 1, 3, 5, and 10 years. For Danish patients, a QoL questionnaire will be distributed electronically, and responses will be automatically integrated into the electronic case report form (eCRF) in REDCap.

Statistical Considerations EuroCUT is designed as a non-inferiority study of KSS ('experimental' arm) compared to RNU ('standard of care' arm) with the primary endpoint of overall survival. The expected 5-year cancer specific mortality after RNU for patients with T0/Ta tumors is 6%. With a 15% mortality due to other causes makes an overall mortality rate of 21% with pT0/pTa tumors. In order to show non-inferiority in patients with a pTa tumor classified as high-risk tumor according to guidelines but imperatively treated with KSS compared to patients who undergo RNU with less than 5% increased risk of overall death, a sample size of 206 patients per arm is required, in order to achieve a power of 80% and a 5% type I error.

Categorical variables will be reported as counts and percentages, and continuous as medians with interquartile range. Test for independence will be performed with the chi-square test for categorical variables and the Wilcox test for numeric variables. Kaplan-Meier, competing-risk and uni- and multivariable COX regression analyses will be applied to assess the probability of recurrence, progression to invasive or metastatic disease, and cancer-specific and overall survival. All tests are planned as two sided with the significance level is set at p < 0.05.

Patient inclusion, data collection and management The recording of data from patient records will be collected prospectively. Primary- or sub-investigators will document updates from the patient records at baseline and follow-up according to the study protocol. No further information will be collected after 10 years, progression to disseminated disease or death.

Data will be reported to the eCRF in the online REDCap web application. The eCRF is stored on a secure server under the responsibility of Zealand University Hospital, Roskilde. REDCap is a secure web application for building and managing online surveys and databases. The study will oblige to the laws and regulations of the Danish Data Protection Agency and EU regulations (GDPR).

All data are kept confidential in a pseudo anonymized form, according to the GDPR and the Danish Data Protection Agency's guidelines. Sponsor will assure that each participant enrolled in the study is coded with a unique patient identification number.

Registry Quality Assurance Measures A structured data dictionary has been developed to align with the eCRF implemented in REDCap. Each variable is defined with a clear name, label, data type (e.g., numeric, categorical, date), permissible values and specified units of measurement where applicable (e.g., serum creatinine in µmol/L).

To ensure data accuracy and consistency, built-in data validation rules are applied within REDCap, including:

* Range checks, used in e.g. height and weight measurement.
* Logic checks (e.g., date of surgery must occur after date of diagnosis etc.)
* Required field enforcement for critical variables
* Conditional branching to prevent irrelevant or contradictory entries throughout the eCRF.
* Format checks (e.g., dates must follow DD-MM-YYYY format) These rules are mirrored in the data dictionary to ensure transparency and traceability. In addition, automated queries are triggered when values fall outside expected ranges or violate logic rules.

The REDCap system is thoroughly tested prior to patient inclusion to ensure reliability and data integrity. A preliminary data extraction has been conducted to confirm that the collected data is suitable for meaningful statistical analysis.

Handling of Missing Data Missing data will be recorded and reported as "Not Available (NA)" in the study dataset and documentation. The primary analyses will be conducted using available data. If the extent or pattern of missing data warrants further consideration, appropriate statistical imputation methods (e.g., multiple imputation) may be employed for selected variables. Any use of imputation will be clearly specified in the statistical analysis plan, and sensitivity analyses will be performed to assess the robustness of the results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed histopathology of UTUC
* Age ≥ 18 years
* Informed patient consent

Exclusion Criteria:

* Patient not willing or able to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with UTUC on a histopatohological specimen from departments of urology within Europe and the USA.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2040-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the end of enrollement until 10 years after inclusion or time of death
  At each follow-up (after 1, 3, 5, and 10 years), we will record whether each participant is alive or has passed away. If a participant has died, we will register whether the cause of death was due to their upper urinary tract cancer or from another cause. This information will be entered into the electronic case report form (eCRF). By doing this, we can better understand how different treatments affect survival related specifically to the cancer.

SECONDARY OUTCOMES:
Cancer specific survival | From the end of enrollement until 10 years after inclusion or time of death
  Cancer specific survival will be assessed by recording the cause of death for all enrolled patients throughout the follow-up period. At each scheduled follow-up time point (1, 3, 5, and 10 years), survival status will be updated, and if applicable, the cause of death will be registered in the electronic case report form (eCRF) as either UTUC-related or due to other causes. This distinction allows for accurate estimation of cancer-specific mortality and evaluation of the oncological safety of different treatment strategies, including kidney-sparing surgery (KSS) versus radical nephroureterectomy (RNU).
Recurrences | From enrollement until five years either after diagnosis or last recurrence according to current follow up guidelines.
  We record the following types of recurrence:
  Any recurrence (local or distant) following radical nephroureterectomy (RNU) or kidney-sparing surgery (KSS).
  Recurrence is documented based on follow-up imaging studies and/or histopathological confirmation.
  Intravesical recurrence following RNU or KSS. All bladder recurrences identified during surveillance cystoscopy are recorded. Additionally, we document any prior or concomitant bladder cancer, in order to differentiate between pre-existing bladder cancer and secondary bladder cancer potentially related to UTUC.
Progression | From enrollment until five years of follow up
  Progression after KSS Progression will be assessed based on histopathological evaluation of local biopsy specimens or subsequent radical nephroureterectomy (RNU) specimens. Both grade progression and stage progression will be recorded according to the WHO 2004/2016 grading system for UTUC.
Renal function | from enrollment until ten years
  Renal function is monitored using serum creatinine (µmol/L) measurements at baseline and at follow-up scheduled at 1, 3, 5, and 10 years. Creatinine values obtained within 3 months prior to each follow-up time point are accepted for analysis.
  The endpoint is the development of chronic kidney disease (CKD) stage ≥3b, defined as an estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m². eGFR is calculated using standard formulas (CKD-EPIkrea), without adjustment for race.
Patient reported outcome measures | Enrollment until five years or death.
  Patient-reported outcomes are assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30). All participants complete the questionnaire at the time of enrollment. Follow-up assessments are administered electronically at 1, 3, and 5 years after inclusion. All responses are included directly into REDCap.

CONTACTS AND LOCATIONS:
Overall Officials: Juan L Vásquez, MD, PhD, Study Director — Zealand University Hospital
Locations (5):
- Denmark (4):
  - Department of Urology Aarhus University Hospital, Aarhus N
  - Herlev Gentofte Hospital, Herlev
  - Department of Urology, Copenhagen University Hospital - Rigshospitalet, København Ø
  - Department of Urology, Zealand University Hospital, Roskilde
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves sensitive personal health information subject to the EU General Data Protection Regulation (GDPR) and Danish data protection laws. These regulations place strict limitations on the disclosure of identifiable or potentially re-identifiable data. As such, IPD will remain confidential and will not be made available to other researchers or third parties outside the approved research team. Summary results will be published in peer-reviewed journals and/or presented at scientific meetings.

REFERENCES:
- [Background] Kealey J, Snider R, Hayne D, Davis ID, Sengupta S. The utility of clinical registries for guiding clinical practice in upper tract urothelial cancer: a narrative review. Transl Androl Urol. 2023 Mar 31;12(3):497-507. doi: 10.21037/tau-22-641. Epub 2023 Mar 16. PMID 37032753
- [Background] Noennig B, Bozorgmehri S, Terry R, Otto B, Su LM, Crispen PL. Evaluation of Intraoperative Versus Postoperative Adjuvant Mitomycin C with Nephroureterectomy for Urothelial Carcinoma of the Upper Urinary Tract. Bladder Cancer. 2018 Oct 29;4(4):389-394. doi: 10.3233/BLC-180174. PMID 30417049
- [Background] Wang Z, Shi H, Xu Y, Fang Y, Song J, Jiang W, Xia D, Wu Z, Wang L. Intravesical Therapy for Upper Urinary Tract Urothelial Carcinoma: A Comprehensive Review. Cancers (Basel). 2023 Oct 17;15(20):5020. doi: 10.3390/cancers15205020. PMID 37894387
- [Background] Erikson MS, Petersen AC, Andersen KK, Jacobsen FK, Mogensen K, Hermann GG. Do repeated transurethral procedures under general anesthesia influence mortality in patients with non-invasive urothelial bladder cancer? A Danish national cohort study. Scand J Urol. 2020 Aug;54(4):281-289. doi: 10.1080/21681805.2020.1782978. Epub 2020 Jun 25. PMID 32584153
- [Background] Seisen T, Granger B, Colin P, Leon P, Utard G, Renard-Penna R, Comperat E, Mozer P, Cussenot O, Shariat SF, Roupret M. A Systematic Review and Meta-analysis of Clinicopathologic Factors Linked to Intravesical Recurrence After Radical Nephroureterectomy to Treat Upper Tract Urothelial Carcinoma. Eur Urol. 2015 Jun;67(6):1122-1133. doi: 10.1016/j.eururo.2014.11.035. Epub 2014 Dec 6. PMID 25488681
- [Background] Raman JD, Ng CK, Boorjian SA, Vaughan ED Jr, Sosa RE, Scherr DS. Bladder cancer after managing upper urinary tract transitional cell carcinoma: predictive factors and pathology. BJU Int. 2005 Nov;96(7):1031-5. doi: 10.1111/j.1464-410X.2005.05804.x. PMID 16225523
- [Background] Lim A, Rao P, Matin SF. Lynch syndrome and urologic malignancies: a contemporary review. Curr Opin Urol. 2019 Jul;29(4):357-363. doi: 10.1097/MOU.0000000000000639. PMID 31045926
- [Background] Rasmussen M, Madsen MG, Therkildsen C. Immunohistochemical Screening of Upper Tract Urothelial Carcinomas for Lynch Syndrome Diagnostics: A Systematic Review. Urology. 2022 Jul;165:44-53. doi: 10.1016/j.urology.2022.02.006. Epub 2022 Feb 22. PMID 35217028
- [Background] Lonati C, Necchi A, Gomez Rivas J, Afferi L, Laukhtina E, Martini A, Ventimiglia E, Colombo R, Gandaglia G, Salonia A, Briganti A, Montorsi F, Mattei A, Simeone C, Carlo MI, Shariat SF, Spiess PE, Moschini M; European Association of Urology Young Academic Urologists EAU-YAU: Urothelial Carcinoma Working Group, the Global Society of Rare Genitourinary Tumors GSRGT. Upper Tract Urothelial Carcinoma in the Lynch Syndrome Tumour Spectrum: A Comprehensive Overview from the European Association of Urology - Young Academic Urologists and the Global Society of Rare Genitourinary Tumors. Eur Urol Oncol. 2022 Feb;5(1):30-41. doi: 10.1016/j.euo.2021.11.001. Epub 2021 Dec 9. PMID 34896051
- [Background] Lonati C, Moschini M, Simeone C, Spiess PE, Necchi A. Lynch syndrome in urological practice: diagnosis, therapeutic strategies, and screening for upper tract urothelial carcinoma. Curr Opin Urol. 2022 Jan 1;32(1):40-47. doi: 10.1097/MOU.0000000000000936. PMID 34608026
- [Background] Tonelli M, Wiebe N, Culleton B, House A, Rabbat C, Fok M, McAlister F, Garg AX. Chronic kidney disease and mortality risk: a systematic review. J Am Soc Nephrol. 2006 Jul;17(7):2034-47. doi: 10.1681/ASN.2005101085. Epub 2006 May 31. PMID 16738019
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Tafuri A, Marchioni M, Cerrato C, Mari A, Tellini R, Odorizzi K, Veccia A, Amparore D, Shakir A, Carbonara U, Panunzio A, Trovato F, Catellani M, Janello LMI, Bianchi L, Novara G, Dal Moro F, Schiavina R, De Lorenzis E, Parma P, Cimino S, De Cobelli O, Maiorino F, Bove P, Crocerossa F, Cantiello F, D'Andrea D, Di Cosmo F, Porpiglia F, Ditonno P, Montanari E, Soria F, Gontero P, Liguori G, Trombetta C, Mantica G, Borghesi M, Terrone C, Del Giudice F, Sciarra A, Galosi A, Moschini M, Shariat SF, Di Nicola M, Minervini A, Ferro M, Cerruto MA, Schips L, Pagliarulo V, Antonelli A. Changes in renal function after nephroureterectomy for upper urinary tract carcinoma: analysis of a large multicenter cohort (Radical Nephroureterectomy Outcomes (RaNeO) Research Consortium). World J Urol. 2022 Nov;40(11):2771-2779. doi: 10.1007/s00345-022-04156-3. Epub 2022 Oct 6. PMID 36203101
- [Background] Hasan MN, Roupret M, Keeley F, Cracco C, Jones R, Straub M, Traxer O, Osther PJS, Brehmer M. Consultation on UTUC, Stockholm 2018 aspects of risk stratification: long-term results and follow-up. World J Urol. 2019 Nov;37(11):2289-2296. doi: 10.1007/s00345-019-02739-1. Epub 2019 Apr 3. PMID 30944969
- [Background] Jung H, Giusti G, Fajkovic H, Herrmann T, Jones R, Straub M, Baard J, Osther PJS, Brehmer M. Consultation on UTUC, Stockholm 2018: aspects of treatment. World J Urol. 2019 Nov;37(11):2279-2287. doi: 10.1007/s00345-019-02811-w. Epub 2019 May 23. PMID 31123852
- [Background] Marcq G, Foerster B, Abufaraj M, Matin SF, Azizi M, Gupta M, Li WM, Seisen T, Clinton T, Xylinas E, Mir MC, Schweitzer D, Mari A, Kimura S, Bandini M, Mathieu R, Ku JH, Guruli G, Grabbert M, Czech AK, Muilwijk T, Pycha A, D'Andrea D, Petros FG, Spiess PE, Bivalacqua T, Wu WJ, Roupret M, Krabbe LM, Hendricksen K, Egawa S, Briganti A, Moschini M, Graffeille V, Autorino R, John P, Heidenreich A, Chlosta P, Joniau S, Soria F, Pierorazio PM, Shariat SF, Kassouf W. Novel Classification for Upper Tract Urothelial Carcinoma to Better Risk-stratify Patients Eligible for Kidney-sparing Strategies: An International Collaborative Study. Eur Urol Focus. 2022 Mar;8(2):491-497. doi: 10.1016/j.euf.2021.03.018. Epub 2021 Mar 26. PMID 33773965
- [Background] Shvero A, Abu-Ghanem Y, Laufer M, Dotan ZA, Zilberman DE, Mor Y, Portnoy O, Fridmen E, Winkler H, Kleinmann N. Endoscopic Treatment for Large Multifocal Upper Tract Urothelial Carcinoma. J Urol. 2021 Apr;205(4):1039-1046. doi: 10.1097/JU.0000000000001505. Epub 2020 Nov 20. PMID 33216692
- [Background] Hendriks N, Baard J, Beerlage HP, Schout BMA, Doherty KSG, Pelger RCM, Kamphuis GM. Survival and Long-term Effects of Kidney-sparing Surgery Versus Radical Nephroureterectomy on Kidney Function in Patients with Upper Urinary Tract Urothelial Carcinoma. Eur Urol Open Sci. 2022 May 2;40:104-111. doi: 10.1016/j.euros.2022.04.007. eCollection 2022 Jun. PMID 35638087
- [Background] Masson-Lecomte A, Birtle A, Pradere B, Capoun O, Comperat E, Dominguez-Escrig JL, Liedberg F, Makaroff L, Mariappan P, Moschini M, Rai BP, van Rhijn BWG, Shariat SF, Smith EJ, Teoh JYC, Soukup V, Wood R, Xylinas EN, Soria F, Seisen T, Gontero P. European Association of Urology Guidelines on Upper Urinary Tract Urothelial Carcinoma: Summary of the 2025 Update. Eur Urol. 2025 Jun;87(6):697-716. doi: 10.1016/j.eururo.2025.02.023. Epub 2025 Mar 20. PMID 40118741
- [Background] Ham WS, Park JS, Jang WS, Kim J. Nephron-Sparing Approaches in Upper Tract Urothelial Carcinoma: Current and Future Strategies. Biomedicines. 2022 Sep 8;10(9):2223. doi: 10.3390/biomedicines10092223. PMID 36140325
- [Background] Soria F, Shariat SF, Lerner SP, Fritsche HM, Rink M, Kassouf W, Spiess PE, Lotan Y, Ye D, Fernandez MI, Kikuchi E, Chade DC, Babjuk M, Grollman AP, Thalmann GN. Epidemiology, diagnosis, preoperative evaluation and prognostic assessment of upper-tract urothelial carcinoma (UTUC). World J Urol. 2017 Mar;35(3):379-387. doi: 10.1007/s00345-016-1928-x. Epub 2016 Sep 7. PMID 27604375
- [Background] Azawi NH, Naeraa SH, Subhi Y, Vasquez JL, Norus T, Dahl C, Thind P, Jensen JB. Oncological outcomes of radical nephroureterectomy for upper urinary tract urothelial neoplasia in Denmark. Scand J Urol. 2020 Feb;54(1):58-64. doi: 10.1080/21681805.2019.1710562. Epub 2020 Jan 16. PMID 31942812
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946